CLINICAL TRIAL: NCT07210762
Title: Gingival Cleft Development at Two Time Points of Canine Retraction: a Split-mouth Randomized Controlled Trial
Brief Title: Gingival Cleft Development at Two Time Points of Canine Retraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Ali Umar, Postgraduate Resident, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUHS-IRB # 174/25
Record Dates: First submitted 2025-08-25; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Gingival Cleft; Orthodontic Space Closure
Keywords: gingival cleft; Orthodontic Space Closure; gingiva; gingival disease; tooth extraction; tooth socket
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Intervention Model Description: split-mouth randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early movement group (Experimental): Canine retraction will be started 1 week after extraction
  Interventions: Other: Early space closure
- Delayed Movement (Experimental): Canine retraction will be started 8 weeks after extraction
  Interventions: Other: Delayed space closure

INTERVENTIONS:
Other: Early space closure — Space closure will be started 1 week after extraction
  Arms: Early movement group
Other: Delayed space closure — Space closure will be started 8 weeks after extraction
  Arms: Delayed Movement

SUMMARY:
The goal of this split-mouth randomized controlled trial is to assess whether the timing of extraction space closure-early vs. delayed initiation-affects the incidence of gingival cleft development in orthodontic patients. The main question it aims to answer is:

Does the incidence of gingival cleft development get influenced by the specific time point at which orthodontic space closure is initiated following extraction?

Quadrants will be assigned to the early movement group and the other to the delayed movement group and extractions will be performed accordingly. These will be assessed for the effect on development of gingival cleft development.

ELIGIBILITY:
Inclusion Criteria:

1. Extraction advised of both first premolars from either maxilla, mandible or both.
2. All permanent dentition present apart from third molars.

Exclusion Criteria:

1. Severe crowding
2. Smokers
3. Patients with systemic diseases that could interfere with bone remodeling.
4. Patients with periodontitis or poor periodontal health.
5. Patients who have previously undergone periodontal surgery in the area of interest.
6. Patients with other oral health conditions that could complicate the treatment or healing process.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
presence of gingival clefts after space closure initiation | start of canine retraction to its completion (approximately 6 months)
  The primary outcome will be the presence of gingival clefts, which will be measured at 3 months and 6 months after space closure initiation

SECONDARY OUTCOMES:
craniofacial growth pattern | craniofacial growth pattern will be measured at baseline
  craniofacial growth pattern from sum of posterior angles
gingival biotype | At baseline (immediately prior to tooth extraction)
  gingival biotype by measuring thickness of gingiva using spreader of size 15
buccal bone dehiscence | Immediately post extraction
  bone dehiscence will be measured utilizing the periodontal probe(in mm) from the distal marginal ridge of premolar as reference point, on both the buccal and palatal/lingual side.
canine bulbosity | will be measured at baseline
  Maximum height of contour of canine will be measured on the pretreatment cast using the digital vernier caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria University of Health Sciences Karachi, Karachi, Sindh, Pakistan